CLINICAL TRIAL: NCT01774942
Title: Effect of Extractions and Straumann Dental Implants on Glycemic Control and Inflammatory Markers in Patients With Diabetes: A Pilot Study
Brief Title: Taking Out All Teeth and Replacing Them With Dentures That Rest on Implants in People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Rahman & Rahman Dental Surgeons, Lahore, Pakistan (Other)
Responsible Party: Principal Investigator, Wenche S. Borgnakke DDS MPH PhD, Adjunct Clinical Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #539-2007; #807_2011; HUM00027142 (Other: University of Michigan Medical School IRB)
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus With Periodontal Complication; Inflammation; Dental Implant Failed
Keywords: Diabetes Mellitus; C-Reactive Protein; Dental Implants, Single-Tooth; Dental Prosthesis, Implant-Supported
MeSH Terms: conditions — Inflammation; Diabetes Mellitus | interventions — Surgical Procedures, Operative; Dental Implants; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Because it is unethical to withhold treatment that is known to be efficacious for severe periodontal infections, there is no control group that would not be treated or that would receive delayed treatment. Enrollment criteria included end-stage ("terminal") periodontal infection of all teeth, which is a condition that must be treated immediately due to its severity and potential for very severe consequences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Procedure/Surgery (Impants/Overdentures) (Experimental): One-arm clinical intervention study: All teeth out, full dentures, dental implants, blood draw. The interventions are not experimental in nature, they are standard procedures, namely extraction of all natural teeth followed by suturing to hold soft tissue in place during initial healing; surgical insertion of commercially available dental implants; and fabrication and re-lining (filling in with acrylic the base of the denture as needed during healing and shrinking of underlying tissue) of full dentures, that is full plates in upper and lower jaw to replace all teeth.
  Interventions: Procedure: Procedure/Surgery

INTERVENTIONS:
Procedure: Procedure/Surgery — All teeth were extracted and replaced by a set of provisional full dentures in upper and lower jaws. Three months after extractions, dental implants were surgically placed and mucosa sutured over them. Three monts later, the dentures were re-lined and fitted onto the implants. Blood draw done by phlebotomist.
  Other Names: All teeth out, full dentures, dental implants, blood draw

SUMMARY:
Gum disease and type 2 diabetes are common chronic diseases that affect each other. Diabetes is increasing, especially in Pakistan. People with diabetes have a greater risk for gum disease. Also, it is thought that that gum disease, a chronic infection, can be a source of systemic inflammation and may contribute to poorer diabetes control.

The aims of this project are to study:

1. Changes in sugar control in people with type 2 diabetes and severe gum disease after having all teeth removed and replaced with Straumann dental implants and full dentures
2. Changes in certain inflammation markers seen with insulin resistance and other diseases and conditions more common in people with diabetes
3. Retention of dental implants in people with type 2 diabetes.

Part I (up to 12 months after implant placement):

The study will recruit 30 patients with type 2 diabetes and severe gum disease from Dr. Amin Rahman's private practices in Pakistan. Their long-term sugar (HbA1c) must be 7.5% or more and the inflammatory marker, C-reactive protein (hsCRP) 1mg/dL or more. Consenting participants will first have an oral examination. Eligible patients will have impressions of the jaws and the color of their teeth and gums recorded. At the next visit, all teeth will be extracted and dentures provided. One week later, there will be a check-up visit. Three months after the teeth were removed, Straumann dental implants will be placed in the jaws. After one week, the patient will be checked again. After three months, the dentures will be adjusted to fit the implants. Follow-up visits will occur every three months until one year after the implants were placed to check the health of the patients as well as their implants, the gums around them, and the dentures. Blood samples will be taken at each follow-up visit.

Part II (from 12 months to 11 years after implant placement):

Follow-up visits will occur every six months for the next ten years, to check the health of the patients as well as their implants, the gums around them, and the dentures. The follow-up visit will be identical to those done in Part I, including blood samples.

DETAILED DESCRIPTION:
Part I:

Our hypotheses are that levels of HbA1c and hsCRP will:

1. decrease after extraction of all teeth
2. not increase after placement of dental implants
3. not increase after prosthetic restoration with full dentures anchored on the dental implants.

Part II:

Our hypothesis is that:

a) the implants will be retained over the long term

Only one arm was included due to ethical reasons: Once potential participants would be diagnosed with terminal periodontal (gum) disease, they would need full-mouth extraction and prosthetic rehabilitation. It would be unethical to withhold or delay treatment that is known to work, especially because such severe gum infection can have very serious consequences. Therefore, no control group was included in study.

Few studies have determined what happens to sugar control and inflammatory markers in people with diabetes if teeth with severe gum disease are removed and replaced with implants and dentures. Neither has any study followed for a total of 11 years after implant placement such subjects that initially had uncontrolled type 2 diabetes as well as recent severe periodontal infection, and several of whom smoke cigarettes.

Therefore, the results of this study could add new understanding about diabetes and dental health. The results of this study could influence dental care guidelines for treating people with uncontrolled or poorly type 2 diabetes and severe gum disease. The option of implant supported dentures could potentially be added to the treatment choices for such patients.

ELIGIBILITY:
Inclusion criteria:

* type 2 diabetes of at least 6 months duration and uncontrolled (HbA1c at least 7.5%)
* all teeth in dentition in need of extraction due to periodontal (gum) disease (end-stage or terminal periodontitis)
* able to return for examination every three months for the first year after implant placement, then every 6 months for five years after implant placement
* willing to have blood drawn at each follow-up visit

Exclusion criteria:

* ≤ 6 natural teeth
* inflammatory conditions/diseases other than type 2 diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2015-08-28 (Actual); Study Completion 2015-08-28 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1a) | Every 3 months/6 months
  Level measured every 3 months during the first year after implant placement; then every 6 months the following 5 years, for a total of 6 years.

SECONDARY OUTCOMES:
high-sensitivity C-reactive protein (hsCRP) | Every 3 months/6 months
  Level measured every 3 months during the first year after implant placement; then every 6 months the following 5 years, for a total of 6 years.

OTHER OUTCOMES:
Retention of implants | 6 years
  Implants sometimes fail if placed in individuals with uncontrolled diabetes, recent infection/inflammation, and cigarette smoking habits. The intent is to evaluate retention of implants in such patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wenche S Borgnakke, DDS MPH PhD, Principal Investigator — University of Michigan; Amin ur Rahman, BDS MPH Cert, Study Director — Rahman & Rahman Dental Surgeons, Lahore, Pakistan; William V Giannobile, DDS MS DMSc, Study Chair — University of Michigan
Locations (1):
- Rahman & Rahman Dental Surgeons, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No